CLINICAL TRIAL: NCT00531297
Title: Endoscopic Posterior Mesorectal Resection in T1 Rectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: Heidelberg University (Other); University of Basel (Other); University of Krakau, Department of Visceral surgery (Unknown)
Responsible Party: Principal Investigator, Ignazio Tarantino, M.D., Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKSG 05/072/2B
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): endoscopic posterior mesorectal resection
  Interventions: Procedure: endoscopic posterior mesorectal resection

INTERVENTIONS:
Procedure: endoscopic posterior mesorectal resection — 6 weeks after local excision of a T1 rectal cancer a rectum sparing endoscopic removal of the dorsal part of the mesorectum by EPMR is performed.

SUMMARY:
Any efforts to spare patients with T1 carcinomas of the rectum from low anterior resection or even abdominoperineal resection are linked to the risk of locoregional recurrence of about 10% (range, 0-24). This is tolerated in the view of the morbidity and mortality risk related to transabdominal resection, which is as high as 7-68% and 0-6.5%, respectively. Accordingly, in addition to transanal local excision various adjuvant therapy schemes with chemo- and/or radiotherapy were developed, given the uncertainty about the lymph node stage. Another approach was to identify histological risk criteria in the primary tumor in terms of defining the limits of rectum-sparing therapy.

In earlier experimental and clinical studies the investigators researched and applied dorsoposterior extraperitoneal pelviscopy, i.e. perineal access to the soft-tissue areas of the minor pelvis using minimally invasive surgery. in T1 carcinoma of the rectum this technique becomes all the more significant, as the perineal approach makes it possible to perform an endoscopic posterior mesorectal resection (EPMR) in combination with rectum-sparing surgery Thereby the relevant lymphatic field of the lower rectum can be removed and histologically examined. As a consequence EPMR should lower the loco-regional recurrence rate, since the most common causes of such are pre-existent but so far not detectable lymph node metastases besides the incomplete resection of the primary tumor.

ELIGIBILITY:
Inclusion Criteria:

* Stage T1 (only)
* Over 18 years old
* Patient's consent
* Previous R0 resection of rectal tumor

Exclusion Criteria:

* Metastases (M1)
* Neoadjuvant chemotherapy or radiotherapy
* Meta- or synchronous tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 5 years

SECONDARY OUTCOMES:
Morbidity (>= CTCAE grade 3) | 30 days
Perioperative mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zerz, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of Surgery, Sankt Gallen, Switzerland